CLINICAL TRIAL: NCT03882632
Title: Evaluation of Fat Grafting Technique Using Autologous Micro-fragmented Autologous Adipose Tissue Lipogems in Fecal Incontinence
Brief Title: Fat Grafting Technique for Fecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Melanie Salerno, RN (Other)
Collaborators: Lifespan (Other)
Responsible Party: Sponsor-Investigator, Melanie Salerno, RN, Dr. Leslie Roth, Brown Physicians, Inc.
Organization: Brown Physicians, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1125611
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Fecal Incontinence (Experimental): Patients will have the opportunity to undergo adipose tissue harvesting and targeted local Injection under ultrasound guidance in muscle defects in the intersphincteric space, all around the remaining portions of the external anal sphincter, and along the course of the pudendal nerves bilaterally
  Interventions: Device: Fat Grafting for Fecal Incontinence

INTERVENTIONS:
Device: Fat Grafting for Fecal Incontinence — Autologous adiopse tissue harvesting/grafting using Lipogems
  Other Names: Fat Grafting

SUMMARY:
Fecal Incontinence affects an estimated 2-20% of the general population, and up to 50% of the elderly and institutionalized population. Patients with incontinence tend to suffer in silence; they often do not seek help because of embarrassment and stigma. They often become confined to their homes because they are afraid of having an "accident". Although this is not a life-threatening condition, the psychological, emotional, and social impact can be devastating.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate reconstructive lipoplasty with micro-fragmented autologous adipose tissue (Lipogems®) in female patients with fecal incontinence. Our hypothesis is that placing approximately up to 90 cc of Lipogems® will yield an effective increase in surviving material (over normal fat injection) due to the refinement of the process and result in decreased fecal incontinence over the long term.

Human Adipose Tissue (Fat) possesses regenerative properties in its stromal vascular fraction (SVF). SVF contains nests of pericytes and human MSC mesenchymal stem cells). MSCs are multipotent cells (also called stromal multipotent cells), that possess the ability to differentiate into various tissues, such as bone, tendon, articular cartilage, ligaments, muscle, and fat. Upon fragmentation of adipose tissue using Lipogems®, viable elements are preserved with pericyte identity within an intact stromal vascular niche. It is hypothesized that upon trauma or disruption of this adipose tissue, the regenerative cells within the intact perivascular niche interact via micro vesicles with the microenvironment at the transplant site to promote angiogenesis, neuronal sprouting and fibroblast production thereby stimulating increased vasculature (circulation, nerve regeneration, muscle growth and tone in the urethral sphincter and in the urethral muscles). If these changes are observed, long lasting regenerative changes occur and should be long lasting versus the shorter live effects of the bulking effect by undisrupted fat tissue.

This is a pilot study of 10 subjects will be treated with local injections of Lipogems® and followed for up to two years. Subjects will receive a full history and examination by a single colorectal surgeon. A clear history of their incontinence frequency, Wexner Incontinence Score, Fecal Incontinence Quality of Life Scale, surgical history, and childbirth history will be collected for all registered patients in order to categorize the study participant according to incontinence-type.

All patients will undergo anal physiology testing and endoanal ultrasound. Pre and post measurements will be recorded and compared for objective evaluation. Patients will be evaluated subjectively with the Wexner incontinence Score and Fecal Incontinence Quality of Life Scale.

Patients will have the opportunity to undergo adipose tissue harvesting and targeted local Injection under ultrasound guidance in muscle defects in the intersphincteric space, all around the remaining portions of the external anal sphincter, and along the course of the pudendal nerves bilaterally. This will be done in the procedure room or operating room with IV sedation and local anesthesia. This will all occur in the same setting on the same day.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >18 < 65 years
2. Sex: females
3. Affected by fecal incontinence (moderate to severe) independently from the etiology and previous treatments
4. No restrictions to follow-up for 24 months after treatment
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Present diagnosis of cancer (not in remission)
2. Patients with uncorrected rectal prolapse
3. Overflow incontinence
4. Patients with neurogenic bowel or spinal cord injuries
5. Any patients unable to give informed consent, including members of vulnerable populations
6. Patients with concomitant pelvic floor disorders, like paradoxical puborectalis contraction or pelvic floor dysfunction
7. Chronic diarrhea
8. Patients with chronic steroid use
9. Patients 17 and under
10. Anal Sepsis (abscess and/or fistula)
11. Inability to undergo the intended diagnostic tests and follow-up
12. Pregnancy
13. Diagnosis of Diabetes Mellitus 1 and 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Patients
Enrollment: 10 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of Fecal Incontinence Measured by patient reported outcomes on questionnaires | 2 years
  Comparison of pre and post procedure outcomes via outcomes questionaires
Resolution of Fecal Incontinence Measured by Physical Exam | 2 years
  Comparison of pre and post procedure outcomes via Endoanal Ultrasound and Physiology Testing

SECONDARY OUTCOMES:
Incident of treatment related adverse events | 2 years
  Site reported adverse events designated as related to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Lifespan, Providence, Rhode Island, United States